CLINICAL TRIAL: NCT06320964
Title: Feasibility and Acceptability of a Group-based Life Skills-integrated Reproductive Health Empowerment Intervention for Newly Married Women, Husbands, and Mothers-in-law
Brief Title: The TARANG Intervention
Acronym: TARANGPilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Collaborators: Network for Engineering and Economics Research and Management (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Vikalp Sansthan (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: R01HD108252_1; R01HD108252 (NIH)
Record Dates: First submitted 2024-03-13; First posted 2024-03-20 (Actual); Results first posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Feasibility; Acceptability; Family Planning; Unintended Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TARANG arm (Experimental): The newly married women received 16 weekly group sessions and one rapport-building session, while the husbands and mothers-in-law received four group sessions each over four months. The TARANG intervention was delivered via gender-matched moderators from Vikalp Sansthan and uses three overarching themes: sexual and reproductive health, gender norms, and empowerment.
  Interventions: Behavioral: TARANG

INTERVENTIONS:
Behavioral: TARANG — For newly married women, the intervention had one introductory rapport-building session, followed by 16 group sessions facilitated by trained female moderators over 5 months. The intervention aimed to empower participants by enhancing their understanding of fundamental topics such as menstruation, conception, and contraception, choice of a method among others. Sessions also covered topics to strengthen participants' sense of agency and their ability to make informed decisions regarding family planning and the timing of their first childbirth. Similarly, for husbands, a male moderator delivered sessions on four topics: Love, Relationships and Expectations; Conception and Health; Contraception Methods, and how to choose family planning methods. For MILs, a female moderator covered four sessions: Nutrition flag, Conception and Health, communication between family members, and the final session on relationships with daughter-in-law.

SUMMARY:
The mixed methods pilot study aims to evaluate the acceptability, feasibility, and implementation challenges of the TARANG intervention in villages in rural/tribal Rajasthan to inform the study design and operational details for a larger cluster-randomized controlled trial.

DETAILED DESCRIPTION:
Participants will participate in the single group in the TARANG intervention arm and receive the sessions that will enable them to navigate newly formed relationships (e.g. spousal communication, healthy relationships with in-laws, establishing peer network, and negotiation skills), improve participants awareness of sexual reproductive health, enable participants to challenge inequitable gender norms to reduce unintended pregnancies.

Newly married women (daughters-in-law) received 17 sessions; husbands received 4 sessions and mothers-in-law received 4 sessions. The sessions are implemented by NGO partner, Vikalp Sansthan via trained facilitators/moderators who are supervised by NGO staff.

In this mixed methods pilot study, we aimed to qualitatively understand the participants' acceptability, feasibility of the TARANG intervention delivery, content, modules, etc. We also aimed to capture the qualitative impact of the TARANG intervention and pilot activities in communities/villages as well as to understand the operational challenges of delivery from participants and NGO moderators (key informants) delivering the intervention. Quantitative pre- and post-surveys were conducted to understand implementation outcomes such as feasibility, acceptability, and satisfaction, among other outcomes.

ELIGIBILITY:
Inclusion Criteria:

Newly married women:

* Age 18-25 years at the time of wedding
* Does not plan to move out of the area for the period of the intervention
* Mother-in-law has agreed to support daughter-in-law's participation in the study
* Mother-in-law and husband are eligible for the study participation

Husbands:

* 18 years or more at the time of the wedding
* Does not plan to move out of the village during period of the intervention
* Mother and wife are eligible for study participation

Mothers-in-law:

* Has a daughter-in-law who is eligible and willing to participate in the study
* Provides individual consent to participate in the study
* Assents for daughter-in-law to participate in the study
* Does not plan to move out of the village during period of the intervention
* The son and the daughter-in-law are eligible for study participation

Exclusion Criteria:

Newly married women:

* Wanting to have a child in the next 12 months at the time of baseline
* Cognitive ability to participate in surveys

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2023-07-14 (Actual); Primary Completion 2024-01-21 (Actual); Study Completion 2024-01-21 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nadia Diamond-Smith, PhD, MS, Principal Investigator — University of California, San Francisco
Locations (1):
- Vikalp Sansthan, Udaipur, Rajasthan, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Gopalakrishnan L, Patil S, Das D, Paul A, Sharma P, Kachhwaha A, Choudhary U, Diamond-Smith N. Feasibility and acceptability of a life skills and reproductive health empowerment intervention for young newly married women in Rajasthan, India: a pre-post convergent mixed methods pilot study. Pilot Feasibility Stud. 2025 Nov 15;11(1):142. doi: 10.1186/s40814-025-01720-7. PMID 41241746
- [Derived] Gopalakrishnan L, Choudhary U, Vallin J, Das D, Sharma P, Kachhwaha A, Panjalingam T, Ruwala R, Diamond-Smith N. Implementation and evaluation of a family planning intervention engaging mothers-in-law of young women in India: a mixed methods pilot study. Glob Health Action. 2025 Dec;18(1):2554435. doi: 10.1080/16549716.2025.2554435. Epub 2025 Sep 8. PMID 40916629
- [Derived] Gopalakrishnan L, Patil S, Das D, Paul A, Sharma P, Kachhwaha A, Choudhary U, Diamond-Smith N. Feasibility and acceptability of a life skills and reproductive health empowerment interventionfor young newly married women in Rajasthan, India: A pre-post convergent mixed methods pilot study. Res Sq [Preprint]. 2024 Oct 16:rs.3.rs-4255712. doi: 10.21203/rs.3.rs-4255712/v1. PMID 39483877
- [Derived] Diamond-Smith N, Vaishnav Y, Choudhary U, Sharma P, Kachhwaha A, Panjalingam T, Vallin J, Das D, Gopalakrishnan L. Individual empowerment and community norm effects of engaging young husbands in reproductive health in rural India: findings from a pilot study. Reprod Health. 2024 Oct 17;21(1):147. doi: 10.1186/s12978-024-01878-y. PMID 39420379
- [Derived] Diamond-Smith N, Vaishnav Y, Choudhary U, Sharma P, Kachhwaha A, Panjalingam T, Vallin J, Das D, Gopalakrishnan L. Individual empowerment and community norm effects of engaging young husbands in reproductive health in rural India: findings from a pilot study. Res Sq [Preprint]. 2024 May 15:rs.3.rs-4376443. doi: 10.21203/rs.3.rs-4376443/v1. PMID 38798481

RESULTS

PARTICIPANT FLOW:
Groups:
- TARANG Arm: Received 16 lifeskills and reproductive health empowerment sessions
Period: Overall Study
Arm/Group | TARANG Arm
Started | 42
Completed | 42
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- TARANG Arm: A single-arm trial in which intervention groups receive an introductory rapport-building session, followed by 16 group sessions facilitated by the moderators over six months. The intervention used practical skill-building activities to empower participants by enhancing their understanding of fundamental topics such as menstruation, conception, and contraception.
Arm/Group | TARANG Arm
Number analyzed (Participants) | 42
Age, Continuous [Mean (Standard Deviation); unit: Years] | 20.3 (1.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 42
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 42
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of the Intervention
Description: Proportion of participants who complete 50% of the intervention sessions
Time Frame: Post-intervention at 5 month endline survey
Population: The outcome was only analyzed for those participants who attended at least one session.
Measure: Count of Participants; unit: Participants
Arm/Group | TARANG Arm
Number analyzed (Participants) | 35
Participants | 28

2. Primary Outcome: Acceptability
Description: Proportion of participants who were completely or somewhat satisfied with the intervention
Time Frame: Post-intervention at 5 month endline survey
Population: Only participants who attended at least one session were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | TARANG Arm
Number analyzed (Participants) | 35
Participants | 34

3. Primary Outcome: Usefulness
Description: Proportion of participants who found the TARANG intervention sessions very useful or somewhat useful
Time Frame: Post-intervention at 5 month endline survey
Population: Only those who attended at least one session were asked about usefulness of sessions.
Measure: Count of Participants; unit: Participants
Arm/Group | TARANG Arm
Number analyzed (Participants) | 35
Participants | 35

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | TARANG Arm
All-Cause Mortality (participants affected / at risk) | 0/42
Serious Adverse Events (participants affected / at risk) | 0/42
Other Adverse Events (participants affected / at risk) | 0/42

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-10-02): https://cdn.clinicaltrials.gov/large-docs/64/NCT06320964/Prot_SAP_ICF_000.pdf